CLINICAL TRIAL: NCT07256964
Title: A Prospective, Randomized Controlled, Multicenter Phase II Clinical Study of Toripalimab Combined With PCb-EC Regimen (Albumin Paclitaxel + Carboplatin Followed by Epirubicin + Cyclophosphamide) or PCb Regimen (Albumin Paclitaxel + Carboplatin) as Neoadjuvant Therapy for Triple-Negative Breast Cancer
Brief Title: Toripalimab Combined With Anthracycline-free or Anthracycline-containing Chemotherapy as Neoadjuvant Chemotherapy for Early Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-TRIO-TORI
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: PD1; TNBC; Neoadjuvant chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCb-EC+PD1 (Active Comparator)
  Interventions: Drug: Toripalimab; Drug: PCb-EC
- PCb+PD1 (Experimental)
  Interventions: Drug: Toripalimab; Drug: PCb

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg every cycle
Drug: PCb-EC — Albumin Paclitaxel + Carboplatin*4 Followed by Epirubicin + Cyclophosphamide*4
  Arms: PCb-EC+PD1
Drug: PCb — Albumin Paclitaxel + Carboplatin *6
  Arms: PCb+PD1

SUMMARY:
This study aims to evaluate the efficacy and safety of a PD-1 inhibitor combined with different chemotherapy regimens (PCb-EC and PCb), in order to develop a superior and well-tolerated neoadjuvant therapeutic strategy for patients with triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years.
2. Disease Status: Clinical pathological confirmation of cT2-cT4d, or cT1c with axillary lymph node metastasis.
3. Pathology: Histopathologically confirmed triple-negative, invasive breast carcinoma.
4. Definition of Triple-Negative Breast Cancer:
5. ER and PR negative (IHC nuclear staining <10%).
6. Her-2 negative (IHC 0 or 1+ without FISH, or IHC 2+ with FISH demonstrating no amplification).
7. Measurable Disease: Presence of clinically measurable lesion(s) confirmed by ultrasound, mammography, or optional MRI within 1 month prior to randomization.
8. Adequate Organ and Bone Marrow Function (within 1 month prior to chemotherapy), indicating no contraindications for chemotherapy:
9. Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L
10. Hemoglobin (Hb) ≥ 90 g/L
11. Platelet count (PLT) ≥ 100 × 10⁹/L
12. Total Bilirubin (TBIL) < 1.5 × ULN (Upper Limit of Normal)
13. Serum Creatinine (Cr) < 1.5 × ULN
14. Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) < 1.5 × ULN
15. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 50% as measured by echocardiogram.
16. Pregnancy Status: For women of childbearing potential, a negative serum pregnancy test within 14 days prior to randomization.
17. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1.
18. Informed Consent: Signed informed consent obtained.

Exclusion Criteria:

1. Metastatic Disease: Evidence of metastatic breast cancer. (To exclude metastasis, CT scans of the chest and abdomen, and a bone scan must be performed at any time point from diagnosis to randomization; PET/CT may serve as an alternative imaging modality).
2. Prior Anti-Cancer Therapy: Any prior chemotherapy, endocrine therapy, targeted therapy, or radiotherapy for the current breast cancer.
3. Second Primary Malignancy: Presence of a second primary malignancy, except for:
4. Adequately treated non-melanoma skin carcinoma.
5. Prior Immunotherapy: Previous treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or any other immunomodulatory therapy.
6. Immunodeficiency or Autoimmune Disease: Diagnosed immunodeficiency or active autoimmune disease requiring systemic treatment.
7. Severe Comorbidities: Severe or uncontrolled pulmonary or cardiac disease.
8. Active Hepatitis: Active Hepatitis B or Hepatitis C infection.
9. Transplantation History: History of solid organ or bone marrow transplantation.
10. Pregnancy/Lactation: Pregnant or lactating women.
11. Other Medical Conditions: Any other severe, uncontrolled medical condition that, in the investigator's judgment, constitutes a contraindication to chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-11-26 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rates | Up to 180 days

SECONDARY OUTCOMES:
Objective response rate（ORR） | up to 180 days
Event-free survival (EFS) | up to 5 years
Invasive Disease-Free Survival (IDFS) | up to 5 years
Overall Survival (OS) | up to 5 years
Adverse events | up to 18 months
EORTC QLQ-C30 questionnaire | up to 18 months
  All of the scales and single-item measures range in score from 0 to 100. A high scale scorerepresents a higher response level
EORTC QLQ-BR23 questionnaire | up to 18 months
  All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning,

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results of the study will be made avaliable after de-indentification.
Time Frame: Within 18 months after the publication of the results.
Access Criteria: Researchers can gain access to the data from the corresponding author upon written request with detailed study plan.